CLINICAL TRIAL: NCT02732639
Title: Open-label, Multicenter, Trial Evaluating Efficacy and Safety of Peginterferon Alfa-2a (PEGASYS®) in Patients With Chronic Hepatitis D (CHD)
Brief Title: A Study of Pegylated Interferon (PEG-IFN) Alfa-2a (Pegasys) in Participants With Chronic Hepatitis D (CHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18788
Record Dates: First submitted 2016-04-05; First posted 2016-04-08 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis D, Chronic
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Pegylated Interferon (PEG-IFN) alfa-2a (Experimental): Participants received pegylated interferon (PEG-IFN) alfa-2a monotherapy for 48 weeks, followed by 24 weeks of treatment-free follow-up.
  Interventions: Drug: Pegylated Interferon (PEG-IFN) alfa-2a

INTERVENTIONS:
Drug: Pegylated Interferon (PEG-IFN) alfa-2a — Participants received pegylated interferon (PEG-IFN) alfa-2a 180 microgram (mcg) subcutaneously (SC) weekly for 48 weeks.
  Other Names: PEGASYS

SUMMARY:
This study evaluated the efficacy and safety of 48-week treatment with pegylated interferon (PEG-IFN) alfa-2a (Pegasys) monotherapy in participants with chronic hepatitis D (CHD). Treatment was followed by 24 weeks of treatment-free follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Positive hepatitis B surface antigen (HBsAg) for at least 6 months prior to screening
* Positive anti-delta for at least 3 months prior to screening
* Positive hepatitis D virus (HDV) ribonucleic acid (RNA)
* A liver biopsy obtained within the past 18 months for non-cirrhotic patients and 30 months for cirrhotic patients demonstrating liver disease consistent with chronic hepatitis D (CHD)
* Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug

Exclusion Criteria:

* Antiviral therapy for CHD within the previous 6 months
* Positive hepatitis A, hepatitis C, or human immunodeficiency virus (HIV)
* Evidence of decompensated liver disease
* Other medical condition associated with chronic liver disease
* Women with ongoing pregnancy or who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Romania (6):
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Craiova
  - Iași
  - Timișoara

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Started | 31
Completed | 30
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Normal Alanine Aminotransferase (ALT) at Week 72
Description: Samples were collected and analyzed for ALT. A normal ALT is a value within the normal range of the assay.
Time Frame: At Week 72
Population: Intention-to-treat (ITT) analysis population included all participants, who received at least one dose of the study medication and had a subsequent post baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
percentage of participants | 54.84 [37.3 to 72.4]

2. Primary Outcome: Percentage of Participants With Negative Hepatitis D Virus Ribonucleic Acid (HDV RNA) at Week 72
Description: Samples were collected and analyzed for HDV RNA levels. Negative HDV RNA is defined as below the level of detection of the assay.
Time Frame: At Week 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
percentage of participants | 61.29 [44.1 to 78.4]

3. Secondary Outcome: Percentage of Participants With Normal ALT at Week 48
Description: Samples were collected and analyzed for ALT levels. A normal ALT is a value within the normal range of the assay.
Time Frame: At Week 48
Population: ITT analysis population included all participants, who received at least one dose of the study medication and had a subsequent post baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
percentage of participants | 45.16 [27.6 to 62.7]

4. Secondary Outcome: Percentage of Participants With Negative HDV RNA at Week 48
Description: as for outcome 2
Time Frame: At Week 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
percentage of participants | 64.52 [47.7 to 81.4]

5. Secondary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Below 1*10^5 Copies/Milliliter (mL) at Weeks 48 and 72
Description: Samples were collected and analyzed for HBV DNA levels. Reported here is the percentage of participants with HBV DNA levels below 1*10^5 copies/mL.
Time Frame: At Weeks 48 and 72
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
percentage of participants
  HBV-DNA at Week 48 | 83.87 [70.9 to 96.8]
  HBV-DNA at Week 72 | 74.19 [58.8 to 89.6]

6. Secondary Outcome: Number of Participants With Positive Hepatitis B Surface Antigen (HBsAg) Levels
Description: Samples were collected and analyzed for HBsAg. Positive HBsAg levels are defined as levels above the level of detection of the assay.
Time Frame: At Screening and at Weeks 48 and 72
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
participants
  HBsAg Positive at Screening | 31
  HBsAg Positive at Week 48 | 29
  HBsAg Positive at Week 72 | 26

7. Secondary Outcome: Percentage of Participants With HBsAg Seronegative at Weeks 48 and 72
Description: Samples were collected and analyzed for HBsAg. Seronegative HBsAg is defined as below the level of detection of the assay.
Time Frame: At Weeks 48 and 72
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
percentage of participants
  Seronegative HBsAg at Week 48 | 0 [NA to NA] — NA: Not applicable since 0% of participants had negative HBsAg measurements.
  Seronegative HBsAg at Week 72 | 3.23 [0.0 to 9.4]

8. Secondary Outcome: Percentage of Participants With Positive Hepatitis B Surface Antibody (HBsAb) at Weeks 48 and 72
Description: Samples were collected and analyzed for HBsAb. Positive HBsAb levels are defined as levels above the level of detection of the assay and reflect the presence of antibodies produced against HBsAg.
Time Frame: At Weeks 48 and 72
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Number analyzed (Participants) | 31
percentage of participants
  Positive HBsAb at Week 48 | 3.23 [0.0 to 9.4]
  Positive HBsAb at Week 72 | 3.23 [0.0 to 9.4]

ADVERSE EVENTS:
Time Frame: Up to week 72
Description: The following adverse events (AEs) were recorded in this study: flu-like symptoms, myalgia, asthenia, headache, weight loss, skin rash, hyperthyroidism, conjunctivitis, neutropenia and thrombocytopenia. Neutropenia and thrombocytopenia were the most frequent AEs. Data to assign numbers to these events are not accessible and therefore not reported.
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights